CLINICAL TRIAL: NCT00480779
Title: Screening, Training, Education and Prevention Service of the University of Pittsburgh, Phase 2
Brief Title: Evaluation of Group Lifestyle Balance DVD in Primary Care Practice
Acronym: STEPUP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Trevor J. Orchard, Professor, University of Pittsburgh
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: W81XWH-04-2-0030
Record Dates: First submitted 2007-05-29; First posted 2007-05-31 (Estimated); Results first posted 2016-06-28 (Estimated); Last update posted 2016-06-28 (Estimated); Status verified 2016-05

CONDITIONS: Prediabetes; Metabolic Syndrome
Keywords: Prediabetes; Metabolic syndrome; Prevention; Lifestyle intervention
MeSH Terms: conditions — Prediabetic State; Metabolic Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- GLB Group (Other): The Group Lifestyle Balance program is a direct adaptation of the Diabetes Prevention Program lifestyle intervention. Participants in the study choose traditional GLB face-to-face group delivery or delivery via DVD. Group members met weekly and completed the program over a 12-15 week period. The face-to-face group meetings were led by a trained lifestyle coach, and participants were encouraged to self-monitor their eating and physical activity behaviors. Participants in both intervention delivery modes received a GLB workbook, fat and calorie counter, pedometer, and self-monitoring books for tracking food intake and physical activity.
  Interventions: Behavioral: GLB Group
- GLB DVD (Other): The Group Lifestyle Balance program is a direct adaptation of the Diabetes Prevention Program lifestyle intervention. Participants in the study choose traditional GLB face-to-face group delivery or delivery via DVD. Those who took part via DVD received an overview of the GLB program at the first session, as well as the materials needed for the program. They subsequently watched one session of the program each week, and received a telephone call from a trained lifestyle coach each week to review weight, physical activity minutes and questions/concerns regarding the program. Participants in both intervention delivery modes received a GLB workbook, fat and calorie counter, pedometer, and self-monitoring books for tracking food intake and physical activity.
  Interventions: Behavioral: GLB DVD

INTERVENTIONS:
Behavioral: GLB Group — The Group Lifestyle Balance (GLB) program is a lifestyle change program adapted from the successful lifestyle intervention utilized in the Diabetes Prevention Program. For this arm, the intervention is delivered in face-to-face groups by a trained lifestyle coach.
  Arms: GLB Group
Behavioral: GLB DVD — The Group Lifestyle Balance (GLB) program is a lifestyle change program adapted from the successful lifestyle intervention utilized in the Diabetes Prevention Program. For this arm, the intervention is delivered via DVD and weekly telephone contact with a trained lifestyle coach.
  Arms: GLB DVD

SUMMARY:
The purpose of this study is to examine different methods of delivering the Group Lifestyle Balance (GLB) intervention (1). The GLB is a 12-week lifestyle change program based on the highly successful lifestyle program that was used in the Diabetes Prevention Program (DPP)(2). A DVD of the Group Lifestyle Program has been developed. Conditions called metabolic syndrome and pre-diabetes increase the risk of diabetes and heart disease. Recent research has shown that type 2 diabetes and metabolic syndrome may be prevented or delayed by making lifestyle changes. A primary care practice will enroll participants who will choose either the GLB-DVD intervention or face-to-face group delivery. Approximately 25 patients will be recruited in each group. It is not known if the GLB intervention delivered via DVD is similarly effective to face-to-face group delivery for people with metabolic syndrome or pre-diabetes. It is hoped that this research study will provide information to help answer that question.

DETAILED DESCRIPTION:
The Group Lifestyle Balance program is a 12-session lifestyle intervention with the same goals for weight loss and physical activity as the successful Diabetes Prevention Program (DPP) lifestyle intervention and has been evaluated in several settings. The DPSC collaborated with the US Air Force Center of Excellence for Medical Multimedia to create a DVD of the GLB. The GLB-DVD is a series of taped sessions of a staged group following a script that was developed to closely follow the program.

Effectiveness was assessed for the intervention delivered via DVD (GLB-DVD) as well as traditionally in a group setting (GLB-GROUP). For each delivery mode, pre- and 3 month post-intervention measures of weight and the achievement of the program goals were assessed. Secondary outcomes measured included assessment of components of the metabolic syndrome (NCEP ATP III) and HbA1c.

The prevention professionals in the practice and the Diabetes Prevention Support Center (DPSC) who provided support for the GLB-DVD and GLB-GROUP participants were health care professionals trained in delivery of the GLB by the DPSC faculty. Group delivery of the GLB was conducted via weekly in person, meetings delivered over 12-15 weeks. For GLB-DVD delivery, an overview of the GLB-DVD and materials was provided at commencement of the intervention. Participants were instructed to view one session/week. At the end of each month the participant was asked to return their DVD via postage-paid mail to the DPSC and the next sequential DVD was mailed to the participant. During GLB-DVD delivery, the DPSC prevention professional contacted the participant weekly via telephone to review weight, physical activity minutes, and questions/concerns regarding the program. Thus, participants in both GLB-GROUP and GLB-DVD were offered a total of 12 health care professional contacts. Participants in both intervention delivery modes received a GLB workbook, fat and calorie counter, pedometer, and self-monitoring books for tracking food intake and physical activity.

ELIGIBILITY:
Inclusion criteria:

* All non-diabetic patients age 18 years and older at the time of enrollment considered to be patients of the practices that are taking part in this project will be eligible for the study upon referral from their physician.
* Non-diabetic patients with metabolic syndrome AND/OR pre-diabetes are eligible for the study with referral from their physician based on the following criteria:

  * Metabolic Syndrome: Patients with BMI greater than or equal to 25 kg/m2, with at least 3 of the following risk factors for metabolic syndrome:

    * Waist circumference (>40 inches men, >35 inches women)
    * Blood pressure greater than or equal to 130 mmHg (systolic) and/or 85 mmHg (diastolic) OR history of diagnosed hypertension
    * Low HDL level (<40mg/dL men, <50 mg/dL women)
    * Elevated triglyceride level greater than or equal to 150 mg/dL
    * Fasting glucose greater than or equal to 100mg/dL and <126mg/dL
  * Pre-diabetes: Patients with a BMI greater than or equal to 25 kg/m2 and pre-diabetes (fasting glucose greater than or equal to 100 mg/dL and <126mg/dL)
* All measures should have been taken within six months of enrollment into the study. The physician in each center will be asked to refer eligible patients to the study. It will be the responsibility of the referring physician to determine eligibility and appropriateness of the patient's participation.

Exclusion Criteria:

* Those patients age less than 18 years old will not be invited to be part of the study. In addition, patients with any of the following conditions are not eligible to take part in the study:

  * Those with previous diabetes diagnosis
  * Women who are currently (or within past 6-weeks) pregnant or lactating
  * Any patient deemed by their physician not to be a candidate
  * Any patient planning to leave the area before the end of the program
  * Individuals that are not patients of the participating primary care practices

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2007-06; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Trevor J Orchard, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Knowler WC, Barrett-Connor E, Fowler SE, Hamman RF, Lachin JM, Walker EA, Nathan DM; Diabetes Prevention Program Research Group. Reduction in the incidence of type 2 diabetes with lifestyle intervention or metformin. N Engl J Med. 2002 Feb 7;346(6):393-403. doi: 10.1056/NEJMoa012512. PMID 11832527
- [Background] Kramer, MK, Miller, R, Venditti, E, Orchard, TO. Group Lifestyle Intervention for Diabetes Prevention in Those with Metabolic Syndrome in Primary Care Practice. Diabetes. June, 2006. 55: Supp., A517.
- See also: Diabetes Prevention Support Center of the University of Pittsburgh — http://www.diabetesprevention.pitt.edu
- See also: A novel approach to diabetes prevention: evaluation of the Group Lifestyle Balance program delivered via DVD — http://www.ncbi.nlm.nih.gov/pubmed/20863586

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients meeting the criteria for participation were referred by their health care provider, who also provided approval for moderate intensity physical activity. After completing informed consent, participants chose which mode of delivery they preferred, GLB-DVD or GLB-GROUP.
Groups:
- GLB Group: The Group Lifestyle Balance program is a direct adaptation of the Diabetes Prevention Program lifestyle intervention. Participants in the study chose traditional GLB face-to-face group delivery or delivery via DVD. Group members met weekly and completed the program over a 12-15 week period. The face-to-face group meetings were led by a trained lifestyle coach, and participants were encouraged to self-monitor their eating and physical activity behaviors. Participants in both intervention delivery modes received a GLB workbook, fat and calorie counter, pedometer, and self-monitoring books for tracking food intake and physical activity.
- GLB DVD: The Group Lifestyle Balance program is a direct adaptation of the Diabetes Prevention Program lifestyle intervention. Participants in the study chose traditional GLB face-to-face group delivery or delivery via DVD. Those who took part via DVD received an overview of the GLB program at the first session, as well as the materials needed for the program. They subsequently watched one session of the program each week, and received a telephone call from a trained lifestyle coach each week to review weight, physical activity minutes and questions/concerns regarding the program. Participants in both intervention delivery modes received a GLB workbook, fat and calorie counter, pedometer, and self-monitoring books for tracking food intake and physical activity.
Period: Overall Study
Arm/Group | GLB Group | GLB DVD
Started | 26 | 22
Completed | 24 | 19
Not Completed | 2 | 3
Not completed — Other | 2 | 0
Not completed — Job and Health-related | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GLB Group | GLB DVD | Total
Number analyzed (Participants) | 26 | 22 | 48
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.0 (11.9) | 57.3 (13.6) | 59.1 (12.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 13 | 34
  Male | 5 | 9 | 14
Region of Enrollment [Number; unit: participants]
  United States | 26 | 22 | 48

OUTCOME MEASURES:

1. Primary Outcome: Change in Weight
Description: The primary outcome for this study will be change in weight measured pre and post intervention.
Time Frame: Baseline and 3 months
Population: Intent to treat using Last Observation Carried Forward (LOCF)
Measure: Mean (Standard Deviation); unit: pounds
Groups:
- GLB DVD: The Group Lifestyle Balance program is a direct adaptation of the Diabetes Prevention Program lifestyle intervention. Participants in the study choose traditional GLB face-to-face group delivery or delivery via DVD. Those who took part via DVD received an overview of the GLB program at the first session, as well as the materials needed for the program. They subsequently watched one session of the program each week, and received a telephone call from a trained lifestyle coach each week to review weight, physical activity minutes and questions/concerns regarding the program. Participants in both intervention delivery modes received a GLB workbook, fat and calorie counter, pedometer, and self-monitoring books for tracking food intake and physical activity.
  GLB DVD: The Group Lifestyle Balance (GLB) program is a lifestyle change program adapted from the successful lifestyle intervention utilized in the Diabetes Prevention Program. For this arm, the intervention is delivered via DVD and
Arm/Group | GLB Group | GLB DVD
Number analyzed (Participants) | 26 | 22
pounds | -13.9 (14.3) | -11.8 (11.4)

2. Secondary Outcome: Change in Waist Circumference
Description: A secondary outcome for this study will be change in waist circumference, measured pre and post intervention.
Time Frame: Baseline and 3 months
Population: Intent to treat
Measure: Mean (Standard Deviation); unit: inches
Arm/Group | GLB Group | GLB DVD
Number analyzed (Participants) | 26 | 22
inches | -2.49 (2.08) | -1.87 (1.98)

3. Secondary Outcome: Change in Total Cholesterol
Description: A secondary outcome for this study will be change in total cholesterol, measured pre and post intervention.
Time Frame: Baseline and 3 months
Population: Intent to treat. Participants with relevant medication changes between baseline and 3 months were excluded.
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | GLB Group | GLB DVD
Number analyzed (Participants) | 24 | 18
mg/dl | -8.29 (27.09) | -9.94 (19.08)

4. Secondary Outcome: Change in HDL Cholesterol
Description: A secondary outcome for this study will be change in HDL cholesterol, measured pre and post intervention.
Time Frame: Baseline and 3 months
Population: Intent to treat. Participants with relevant medication changes between baseline and 3 months were excluded.
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | GLB Group | GLB DVD
Number analyzed (Participants) | 24 | 18
mg/dl | -2.08 (5.9) | -0.72 (3.71)

5. Secondary Outcome: Change in LDL Cholesterol
Description: A secondary outcome for this study will be change in LDL cholesterol, measured pre and post intervention.
Time Frame: Baseline and 3 months
Population: Intent to treat. Participants with relevant medication changes between baseline and 3 months were excluded.
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | GLB Group | GLB DVD
Number analyzed (Participants) | 24 | 18
mg/dl | 0.33 (20.87) | -2.67 (14.69)

6. Secondary Outcome: Change in Fasting Glucose
Description: A secondary outcome for this study will be change in fasting glucose, measured pre and post intervention.
Time Frame: Baseline and 3 months
Population: Intent to treat. Participants with relevant medication changes between baseline and 3 months were excluded.
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | GLB Group | GLB DVD
Number analyzed (Participants) | 26 | 21
mg/dl | 1.15 (10.52) | -4.71 (6.66)

7. Secondary Outcome: Change in Hemoglobin A1C
Description: A secondary outcome for this study will be change in HbA1c, measured pre and post intervention. The hemoglobin HbA1c test provides information regarding how well blood glucose (sugar) has been controlled for the previous 8-12 weeks..
Time Frame: Baseline and 3 months
Population: Intent to treat. Participants with relevant medication changes between baseline and 3 months were excluded.
Measure: Mean (Standard Deviation); unit: percentage of glycosylated hemoglobin
Arm/Group | GLB Group | GLB DVD
Number analyzed (Participants) | 26 | 21
percentage of glycosylated hemoglobin | -0.31 (0.25) | -0.16 (0.23)

8. Secondary Outcome: Change in Systolic Blood Pressure
Description: A secondary outcome for this study will be change in systolic blood pressure, measured pre and post intervention.
Time Frame: Baseline and 3 months
Population: Intent to treat. Participants with relevant medication changes between baseline and 3 months were excluded.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | GLB Group | GLB DVD
Number analyzed (Participants) | 20 | 21
mmHg | -6.55 (11.29) | -4.95 (6.68)

9. Secondary Outcome: Change in Diastolic Blood Pressure
Description: A secondary outcome for this study will be change in diastolic blood pressure, measured pre and post intervention.
Time Frame: Baseline and 3 months
Population: Intent to treat. Participants with relevant medication changes between baseline and 3 months were excluded.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | GLB Group | GLB DVD
Number analyzed (Participants) | 20 | 21
mmHg | -3.6 (7.68) | -1.43 (6.88)

10. Secondary Outcome: Change in Triglycerides
Description: A secondary outcome for this study will be change in Triglyceride level, measured pre and post intervention.
Time Frame: Baseline and 3 months
Population: Intent to treat. Participants with relevant medication changes between baseline and 3 months were excluded.
Measure: Median (Inter-Quartile Range); unit: mg/dl
Arm/Group | GLB Group | GLB DVD
Number analyzed (Participants) | 26 | 22
mg/dl | -2.0 [-43 to 1] | 0 [-26 to 0]

ADVERSE EVENTS:
Groups:
- GLB DVD: The Group Lifestyle Balance program is a direct adaptation of the Diabetes Prevention Program lifestyle intervention. Participants in the study choose traditional GLB face-to-face group delivery or delivery via DVD. Those who took part via DVD received an overview of the GLB program at the first session, as well as the materials needed for the program. They subsequently watched one session of the program each week, and received a telephone call from a trained lifestyle coach each week to review weight, physical activity minutes and questions/concerns regarding the program. Participants in both intervention delivery modes received a GLB workbook, fat and calorie counter, pedometer, and self-monitoring books for tracking food intake and physical activity.
  GLB DVD:The Group Lifestyle Balance (GLB) program is a lifestyle change program adapted from the successful lifestyle intervention utilized in the Diabetes Prevention Program. For this arm, the intervention is delivered via DVD and
Arm/Group | GLB Group | GLB DVD
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/22
Other Adverse Events (participants affected / at risk) | 0/26 | 0/22

LIMITATIONS AND CAVEATS:
It should be noted that this was a small pilot study and should be tested in a larger sample.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No